CLINICAL TRIAL: NCT00326378
Title: A Multinational, Multicenter, Phase III Open Randomized Trial With or Without Consolidation Chemotherapy Using Docetaxel and Cisplatin After Concurrent Chemoradiation in Inoperable Stage III Non-small Cell Lung Cancer (CCheIN)
Brief Title: Efficacy Study of Additional Chemotherapy After Concurrent Chemoradiation in Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Keunchil Park, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-08-066
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2012-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Consolidation Chemotherapy; Docetaxel; Cisplatin

ARMS (2):
- CCRT arm without consolidation chemotherapy (Active Comparator): Docetaxel 20mg/m2 & Cisplatin 20mg/m2 (D1,8,15,22,29,36) during radiotherapy
  Interventions: Drug: CCRT arm without consolidation chemotherapy
- CCRT arm with consolidation chemotherapy (Experimental): docetaxel 20mg/m2 & cisplatin 20mg/m2 (D1,8,15,22,29,36) during radiotherapy, and followed by consolidation chemotherapy with 3-weekly docetaxel 35mg/m2 & cisplatin 35mg/m2 (D1,8) every 3 weeks (#3).
  Interventions: Drug: consolidation chemotherapy with Docetaxel plus cisplatin

INTERVENTIONS:
Drug: consolidation chemotherapy with Docetaxel plus cisplatin — definitive CCRT, and followed by consolidation chemotherapy with three cycles of docetaxel plus cisplatin
  Arms: CCRT arm with consolidation chemotherapy
Drug: CCRT arm without consolidation chemotherapy — definitive CCRT with weekly Docetaxel/CDDP #6 without consolidation chemotherapy
  Arms: CCRT arm without consolidation chemotherapy

SUMMARY:
Non-Small Cell Lung Cancer(NSCLC) is the leading cause of death in Korean men after stomach cancer. Surgical resection plays a main role for curative treatment. However, less than 20 % of the NSCLC patients have been found in stage I-II disease. In inoperable stage IIIA/B disease, the recommended treatment is combined chemotherapy and radiation therapy. Various kinds of combination of 2 modalities have been used either in sequential or concurrent setting. Concurrent chemoradiotherapy(CCRT) have been recognized to have better survival than radiation therapy alone or sequential therapy, but additional consolidation chemotherapy after CCRT is not yet to be determined for the beneficial role in survival gain. Docetaxel is an anticancer drug and has synergistic anticancer effect in various cancer with cisplatin, another anticancer drug. In the present study, randomised trial will be performed to confirm the efficacy of the consolidation chemotherapy with docetaxel and cisplatin after completing CCRT with the same chemotherapeutic agents in stage III inoperable NSCLC on progression free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small cell lung cancer
* Presence of measurable disease by RECIST
* Inoperable Stage IIIA or IIIB, proven by CT or MRI (except wet T4). However, N2 or N3 should be confirmed by PET or pathology. (For T4, PET is optional)
* 18 years of age or older
* ECOG Performance status 0-1
* No prior chemotherapy, radiation therapy to chest, immunotherapy, or biologic therapy
* Serum Hgb ≥ 10 gm/dL, platelet ≥ 100,000/μL, absolute neutrophil count ≥ 1,500/μL
* Serum creatinine ≤1.25 x UNL or creatinine clearance ≥60 mlmL/min
* Serum bilirubin ≤ 1.5 x UNL, AST (SGOT) and ALT (SGPT) ≤ 2.5 x UNL, alkaline phosphatase ≤ 5 x UNL
* FEV1> 0.8 L
* Patients must sign an informed consent

Exclusion Criteria:

* Carcinoid tumor, small cell carcinoma of lung
* Patients with any distant metastasis
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
* Any other morbidity or situation with contraindication for chemotherapy (e.g. active infection, myocardial infarction preceding 6 months, symptomatic heart disease including unstable angina, congestive heart failure or uncontrolled arrhythmias, immunosuppressive treatment)
* Pregnant or lactating women, women who has not taken test of pregnancy (within 14 days before the first administration) and pregnant women
* Women and men of childbearing potential who have no willing of employing adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2005-10; Primary Completion 2013-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Progression free survival | The final analysis will be conducted when 381 events (progressions or deaths) are observed.

SECONDARY OUTCOMES:
overall survival | The final analysis will be conducted when 381 events (progressions or deaths) are observed.
response rate | The final analysis will be conducted when 381 events (progressions or deaths) are observed.
patterns of failure | The final analysis will be conducted when 381 events (progressions or deaths) are observed.
safety | The final analysis will be conducted when 381 events (progressions or deaths) are observed.

CONTACTS AND LOCATIONS:
Overall Officials: Keunchil Park, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Ahn JS, Ahn YC, Kim JH, Lee CG, Cho EK, Lee KC, Chen M, Kim DW, Kim HK, Min YJ, Kang JH, Choi JH, Kim SW, Zhu G, Wu YL, Kim SR, Lee KH, Song HS, Choi YL, Sun JM, Jung SH, Ahn MJ, Park K. Multinational Randomized Phase III Trial With or Without Consolidation Chemotherapy Using Docetaxel and Cisplatin After Concurrent Chemoradiation in Inoperable Stage III Non-Small-Cell Lung Cancer: KCSG-LU05-04. J Clin Oncol. 2015 Aug 20;33(24):2660-6. doi: 10.1200/JCO.2014.60.0130. Epub 2015 Jul 6. PMID 26150444